CLINICAL TRIAL: NCT04215679
Title: Comparison of Three Dimensional Virtual Reality Therapy and Motor Imaging in Functional Recovery of Upper Extremity After Stroke
Brief Title: Effect of Motor Imagery With Virtual Reality in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-RK-05
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Virtual reality; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The first group of the study is immersive virtual reality therapy (IVR), the second group is motor imagery therapy (MI), and the third group is the conventional physiotherapy group (CG).
Who Masked: Outcomes Assessor
Masking Description: Participant will be evaluated at baseline, 6 weeks later by an another investigator who does not aware of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Three-dimensional immersive virtual reality application (Experimental): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose mini Mental State Examination (MMSE) scores equal or above the 25 will be included in this study. Oculus Rift and Leap motion will be used to create an immersive interactive environment. Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire,Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied just before the rehabilitation program, after the application and at the end of 6 weeks.
  Interventions: Other: Three-dimensional immersive virtual reality application
- Motor imagery (Active Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Oculus Rift and Leap motion will be used to create an immersive interactive environment. Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire,Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied just before the rehabilitation program, after the application and at the end of 6 weeks.
  Interventions: Other: Motor imagery
- Conventional physiotherapy (Active Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Oculus Rift and Leap motion will be used to create an immersive interactive environment. Modified Ashworth Scale (MAS), Functional independence scale, self-care questionnaire,Action Research Arm Test, Fugl meyer upper extremity motor evaluations will be applied just before the rehabilitation program, after the application and at the end of 6 weeks.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Three-dimensional immersive virtual reality application — In this group, individuals will be included in a game program that will last for 3 days a week for a total of 6 weeks and 45 minutes a day. Individuals will use the IVR to rehabilitate functions that are frequently used in daily life through task-oriented games. The IVR device will be placed on the head of the individual by closing the eyes of the individual and the Leap Motion device will be used to enable individuals to see their own hands in a virtual reality environment. In order to ensure the safety of individuals, practices shall be carried out with the individual sitting in the chair and leaning against the back. A total of 3 different games will be used for upper extremity function, each game will be 15 minutes and the total session time will be 45 minutes.
  Arms: Three-dimensional immersive virtual reality application
Other: Motor imagery — Motor imagery will be performed with the eyes closed. In addition, for the safety of the individual, the individual will sit comfortably in a chair in a quiet environment and sit back. In the motor imagery group, individuals will be shown videos of the 3 games for 2 times in the IVR group and will be asked to imagine that they perform the same functions in the IVR games. The motor imagery will be 3 days a week for a total of 6 weeks and 45 minutes per day (including rest periods).
  Arms: Motor imagery
Other: Conventional physiotherapy — Individuals in this group will be randomly recruited from hospitalized stroke volunteers. Since these individuals receive routine rehabilitation 5 days a week, they will be evaluated at the beginning and end of 18 sessions over a total period of 6 weeks. Conventional physiotherapy will include normal joint movements, muscle strengthening exercises, balance and mobility exercises, and exercises to improve daily life activity.
  Arms: Conventional physiotherapy

SUMMARY:
Virtual reality applications in hemiplegia rehabilitation are gaining popularity. It is claimed that, apart from implementing a function, imagining that function can trigger synaptic connections.

DETAILED DESCRIPTION:
Although the effects of non-three-dimensional virtual reality and motor imagination on the brain have been investigated in a study, such comparison has not been made between the three-dimensional virtual reality and motor imagery.

Considering these situations, the aim of this study is to compare the effect of three-dimensional (immersive) virtual reality and motor imagery on upper extremity functional recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as stroke patient.
* Speaks, reads and writes in Turkish.
* Hand functions at 4, 5, 6 levels according to Brunnstrom.
* Mini mental test score to be at least 24.
* Volunteer for participation.

Exclusion Criteria:

* Neurological, orthopedic problems other than stroke.
* To have motion sickness that cannot continue 3D application.
* Individuals neglecting the affected side

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Jebsen Hand Function Test | 6 weeks
  The test consists of 7 subtitles and is an objective and standardized test. The test consists of 7 subtitles: "writing a standard sentence", "flipping 5 cards", "picking up small objects", "feeding simulation", "arranging backgammon checkers", "carrying large light objects" and "carrying large heavy objects". The score of the test is the completion time of the test and is recorded in seconds
Action Reach Arm Test (ARAT) | 6 weeks
  This scale is scored between 0-57 points and consists of 4 headings: gross grip, fine grip, fingertip grip, and gross motion. Each part is calculated over 3 points. 3 points mean that the test is done in a normal way, 2 points show the difficulty and abnormally long time for doing it, 1 point means that individual can partially complete the test and 0 points can not complete the test. The higher the score, the better the level.

SECONDARY OUTCOMES:
Stroke impact scale (SIS) | 6 weeks
  Turkish validity was done by Hantal et al. in 2014. It is a 9-stage scale that is scored between 0-57 points, with a higher score indicating a better condition and a lower score indicating a higher severity of stroke. Scoring is done separately for each title
Kinesthetic and visual imagery questionnaire | 6 weeks
  It was developed in 2007 by Malouin et al. In this method, the participant is told about the desired movement and is asked to do so. Then the participant is asked to imagine as if he was watching the movement without making any movement. It is scored between 1-5 points. 1: no image, 5: as clear as the original. At the other stage, he is asked to imagine himself by feeling what he is doing and is scored between 1 and 5 points. 1 point: no sense, 5 points mean intense feeling as if he is making the move. The scale assesses both visual and kinesthetic imagery with each dimension being scored from 5 to 25 with higher scores indicating greater imagery clarity or intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University; Ramazan KURUL, Ph.D, Principal Investigator — Bolu Abant Izzet Baylsa University; Muhammed Nur Ögün, MD, Principal Investigator — Bolu Abant Izzet Baylsa University; Şebnem AVCI, Ph.D, Study Director — Bolu Abant Izzet Baylsa University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No